CLINICAL TRIAL: NCT06627881
Title: Effect of Three Training Programs on the Cardiovascular Condition of Individuals with Spinal Cord Injury, a Model of Autonomic Nervous System Dysfunction.
Brief Title: Effect of Three Training Programs on the Cardiovascular Condition of Individuals with Spinal Cord Injury
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Instituto Nacional de Rehabilitacion (Other Government)
Responsible Party: Principal Investigator, Marlene Alejandra Rodríguez Barragán, MD, MSc, Instituto Nacional de Rehabilitacion
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 01/24
Record Dates: First submitted 2024-10-03; First posted 2024-10-04 (Actual); Last update posted 2024-10-04 (Actual); Status verified 2024-01

CONDITIONS: Spinal Cord Injuries; Cardiovascular Condition; Exercise
MeSH Terms: conditions — Spinal Cord Injuries; Motor Activity

STUDY DESIGN:
Intervention Model Description: Randomized clinical trial
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Those in charge of evaluating results and the person in charge of statistical analysis will be blinded and will not know the assignment of the intervention. The person in charge of carrying out the assigned exercise and the participant will know the assignment of the intervention.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Continuous aerobic kayak training program (Experimental): * Frequency: 5 days a week.
  * Intensity: moderate 40.59% RHR or Borg 12-13. Progressing 3rd week 60-70% FCR, Borg 14-17.
  * Time: 8 weeks
  * Volume:
    5 min warm up upper body and center of the upper body 30 minutes of training Progression after 3 weeks: 35 min Total of 40 sessions.
  Interventions: Other: Continuous aerobic kayak training program
- Aerobic Endurance Circuit Program (Active Comparator): * Frequency: 5 days a week.
  * Intensity: Very light <30% of 1 RM, Borg <9 Progression in week 3: light 30-40% of 1 RM, Borg 9-11
  * Time: 8 weeks
  * Volume: 30 min 5 min upper body and center warm-up 2 aerobic resistance circuits with 8 upper body and core exercises, 18-22 repetitions Week 3 progression: 3 circuits Week 4 progression: 4 circuits Recovery period between circuits: 3 min Total of 40 sessions.
  Interventions: Other: Aerobic Endurance Circuit Program
- High intensity interval program with rope (Active Comparator): * Frequency: 5 days a week.
  * Intensity: Vigorous <30% of RHR, Borg 14-17 with recovery interval intensity of 30-39% of RHR Borg 9-11
  * Time: 8 weeks
  * Volume: 30 min 5 min upper body and center warm-up Start: 1:3 ratio, intensive intervals lasting 1 min and recovery interval of 3 min, performing 7 intervals with a total duration of 28 min Progression week 3: Interval ratio will be modified 1:2, performing 10 intervals.
  Total of 40 sessions.
  Interventions: Other: High intensity interval program with rope

INTERVENTIONS:
Other: Continuous aerobic kayak training program — Sitting in a special chair on the Kayak Pro® Speed Stroke PRO ergometer. 5-minute warm-up and continuous training, for 30 minutes on the ergometer at a moderate to vigorous intensity, 5 days a week.
  Arms: Continuous aerobic kayak training program
Other: Aerobic Endurance Circuit Program — Sitting with feet flat on the floor and shoulder-width apart, in each session with a 5-minute warm-up, light intensity training with upper body strengthening, 5 days a week.
  Arms: Aerobic Endurance Circuit Program
Other: High intensity interval program with rope — Sitting with feet flat on the floor and shoulder-width apart, in each session with a 5-minute warm-up, vigorous intensity undulating rope training using the interval method, 5 days a week.
  Arms: High intensity interval program with rope

SUMMARY:
Objective: Describe the effect of different aerobic training programs on the autonomic nervous system (ANS), cardiovascular condition, body composition, metabolic profile, movement and functional independence in patients with spinal cord injury (SCI).

Design: Randomized clinical trial Participants: Individuals in the chronic phase of SCI. Interventions: Three training programs: continuous aerobic in kayak, aerobic resistance circuit, and high-intensity interval with rope. The main measures to be explored will be the potential effects of training on heart rate variability as an indicator of autonomic function; measurement of oxygen consumption (VO2max) and resting metabolic unit (METs) for cardiovascular fitness; bone density examination (DXA) for body composition, metabolic profile, functional independence and life satisfaction in individuals with SCI.

Results: The 8-week training program will increase METs and VO2max, improve heart rate variability and anthropometric variables, body composition, and metabolic profile

DETAILED DESCRIPTION:
Background The increased overall cardiovascular risk could have some causes, such as dyslipidemia, diabetes mellitus, hypertension (HTN), higher BMI, higher waist-to-hip ratio, or deterioration in physical fitness. Obesity and diabetes have been shown to be comparatively higher among people with SCI. An additional factor that contributes to the high cardiovascular morbidity and mortality in SCI is sedentary lifestyle and reduced physical function associated with the loss of motor function, and the interruption of normal autonomic cardiovascular control mechanisms.

It is increasingly recognized that inflammation plays an important role in the development of cardiovascular disease (CVD); elevated reactive C protein (RCP) levels are independently associated with increased all-cause mortality, cardiovascular death, and cardiovascular events. In turn, the higher degree of dyslipidemia found in the population with SCI contributes significantly to this risk. Abnormal lipids are generally modifiable with changes in physical activity and diet along with the use of statins. Numerous studies in people with diabetes have unequivocally shown that hyperglycemia is a potent risk marker for CVD; altered carbohydrate metabolism is more common in people with SCI, and is believed to appear at an earlier age than in people without disabilities.

High adiposity and visceral fat accumulation are related to insulin resistance, gluco-metabolic disorders and a higher risk of developing DM (diabetes mellitus) and CVD. Sophisticated and high-precision radiological techniques, such as DXA and CT, are considered the gold standards for accurate measurement of the ratio of lean to fat mass, it is proposed that the increase in body fat mass and the decrease in Lean tissue mass are valuable markers of CVD.

Exercise has been shown to have good results, mainly in the early stages of BF. In particular, it has been described that aerobic exercise training improves baroreflex sensitivity and that the magnitude of the improvement is related to the intensity of the exercise performed and is proportional to the gains in aerobic capacity (through VO2max). However, in advanced stages of CVD, the response to exercise may be affected due to ANS dysfunction. Indeed, autonomic dysfunction plays a primary role in the pathophysiology of coronary ischemic disease. The presence of a high HRV is a sign of good adaptability and implies that the individual has autonomic control mechanisms that function adequately, that is, the activity of this system plays a substantial role in the physiological adaptations of circulation to changes in brain activity. human being. Therefore, the study of pathologies that affect the ANS can help understand this lack of response and search for effective strategies to improve cardiovascular function.

To date, there are few studies that have evaluated the effect of different exercise modalities on the cardiovascular condition of people with SCI, who will have a different response from that of healthy people or at the beginning of chronic diseases, but similar to that of people in advanced stages of cardiovascular disease. Therefore, exercise can exert cardioprotective effects and benefit the cardiovascular risk profile.

Justification:

A SCI is accompanied by alterations in the autonomic nervous system that lead to an increase in cardiovascular risk in the chronic stages (after 6 months of the injury). In view of the high prevalence of cardiovascular disease, health consequences, and costs associated with SCI, greater emphasis should be placed on identifying therapeutic interventions that reduce cardiovascular risk factors.

It is documented that intervention with low to moderate intensity aerobic exercise induces favorable adaptations in patients with chronic SCI and reduces cardiovascular risk.

However, individuals with SCI face physical impairments and psychological barriers that increase the challenge of implementing exercise into their daily lives. Therefore, prescribing and controlling exercise intensity presents its own difficulties, particularly for people with an altered heart rate response to exercise.

Knowing the effect of aerobic exercise in individuals with SCI will allow the implementation of a training program in a timely manner that will help prevent cardiovascular diseases. It will also improve physical fitness levels, which makes it easier to carry out activities of daily living and, in turn, improves quality of life.

The National Rehabilitation Institute is a place of concentration for the care of people with SCI, and each year approximately 250 first-time specialized consultations are granted to people with said diagnosis. In addition, there is a multidisciplinary team and the necessary infrastructure to carry out this project.

Research question:

What is the effect of three different aerobic training programs on cardiac autonomic system, cardiovascular fitness, body composition, metabolic profile, and independence in people with SCI?

Hypothesis:

The 8-week continuous aerobic kayak training program will increase METs and VO2max, improve heart rate variability and anthropometric variables, body composition, metabolic profile, muscle strength, functional independence and life satisfaction significantly compared to aerobic resistance circuit exercise and high-intensity interval rope exercise.

OBJECTIVES to. General objective:

* Describe the effect of 3 different training programs (continuous aerobic in kayak, aerobic resistance circuit and high intensity interval with rope) on the cardiac autonomic system, cardiovascular fitness, body composition, metabolic profile and independence in individuals with injury medullary.
* Describe the correlation between the R-R interval, VO2max, METs and possible correlating factors such as age, NLI, AIS and chronicity of the injury.

Clinical and demographic outcome measurements:

SCI severity: According to American Spinal Injury Association, with International standards for neurological classification of spinal cord injury modifications: complete, B: incomplete, preservation of only the sensitive function, C: incomplete, voluntary anal contraction or more than half of key muscles in <3, D: incomplete, more than half of the key muscles in >3, E: total recuperation A, B, C, D, E Neurological level: More caudal segment of the SC with normal function Time of evolution of the SCI:Time in days elapsed from when the SCI was produced until time of application of the questionnaire Age:Years elapsed from date of birth to time of questionnaire application

SCI severity: According to American Spinal Injury Association, with International standards for neurological classification of spinal cord injury modifications: complete, B: incomplete, preservation of only the sensitive function, C: incomplete, voluntary anal contraction or more than half of key muscles in <3, D: incomplete, more than half of the key muscles in >3, E: total recuperation A, B, C, D, E Neurological level: More caudal segment of the SC with normal function Time of evolution of the SCI:Time in days elapsed from when the SCI was produced until time of application of the questionnaire Age:Years elapsed from date of birth to time of questionnaire application

SCI severity: According to American Spinal Injury Association, with International standards for neurological classification of spinal cord injury modifications: complete, B: incomplete, preservation of only the sensitive function, C: incomplete, voluntary anal contraction or more than half of key muscles in <3, D: incomplete, more than half of the key muscles in >3, E: total recuperation A, B, C, D, E Neurological level: More caudal segment of the SC with normal function Time of evolution of the SCI:Time in days elapsed from when the SCI was produced until time of application of the questionnaire Age:Years elapsed from date of birth to time of questionnaire application

* SCIM III (Spinal Cord Independence Measure) Measurement of Functional Independence in spinal cord injuries
* LiSAT-9 Life Satisfaction Scale
* VO2max Oxygen consumption
* METs Metabolic equivalents
* STD RR Time domain measurement of cardiac variability
* RMSSD Time domain measurement of cardiac variability
* pNN50 Time domain measurement of cardiac variability
* VLF Frequency domain measurement of very low frequency cardiac variability
* LF Frequency domain measurement of low frequency cardiac variability
* HF Frequency domain measurement of high frequency cardiac variability
* LF/HF Frequency domain measurement of cardiac variability
* Serum glucose plasma glucose concentration.
* Triglycerides concentration of triglycerides in plasma.
* HDL cholesterol amount of cholesterol linked to high-density lipoproteins (HDL-C)
* LDL cholesterol amount of cholesterol bound to low-density lipoproteins.
* Serum insulin hormone involved in the regulation of carbohydrate metabolism.
* Ultrasensitive PCR Acute phase reactant that is released in response to inflammatory processes
* total body fat percentage of total body fat
* Android fatty tissue
* Android fat tissue percentage
* Gynecoid fatty tissue Percentage of gynecoid fatty tissue
* A/G ratio Android fat tissue/gynecoid fat tissue ratio
* VAT mass Visceral adipose tissue
* VAT Visceral adipose tissue volume
* VAT visceral adipose tissue area
* Appen. lean/ height Relationship between appendicular lean mass and height (ALM/Height2)
* Body mass index Weight of a person in kilograms divided by the square of height in meters in individuals with BF
* Diet Adherence Percentage of subjects with diet adherence
* Clinical trunk control test Ability to perform different activities related to balance and trunk movement
* Instrumented Trunk Control Test Trunk stability evaluated using inertial measurement units (IMUs)
* Max Torque Ext Maximum force generated by a muscle or muscle group during a concentric contraction in the extension phase of a specific joint
* Torque max Flex Maximum force generated by a muscle or muscle group during a concentric contraction in the flexion phase of a specific joint.
* Maximum power Ext Rate of work done or the amount of energy generated per unit of time in a muscle group during a concentric contraction in the extension phase of a specific joint, in an isokinesia test
* Maximum Flex Power Rate of work performed or the amount of energy generated per unit of time in a muscle group during a concentric contraction in the Flexion phase of a specific joint, in an isokinesia test
* Total Work Ext Amount of energy transferred or performed by a force when applied over a distance during an Extension exercise.
* Total Work Flex Amount of energy transferred or performed by a force when applied over a distance during a Flexion exercise.

DESIGN AND METHODOLOGY Type of study: Randomized clinical trial (RCT). Description of the work universe: Patients from the outpatient clinic and hospitalization of the Spinal Injury service of the National Rehabilitation Institute, with a diagnosis of spinal cord injury of any etiology, any type (complete and incomplete), with neurological level below C8, of more than 6 months of evolution.

Inclusion Criteria.

* Age over 18 years
* Any sex
* Spinal cord injury due to any etiology
* With clinical diagnosis of spinal cord injury of any type (complete and incomplete)
* With a clinical diagnosis of spinal cord injury with a neurological level below C8 (who are able to lift or/and grab the paddle, ropes, resistance bands or weights)
* With evolution time greater than 6 months
* Adequate trunk control (trunk control scale >13 points)
* That you have a letter of informed consent.

Elimination criteria:

• That another cardiovascular pathology be added

Sample size: A previous INRLGII study found an effect size of 12.6 with a standard deviation of 3.6 with kayak ergometer training compared to conventional therapy. With the Epidata 4.2 program, the sample was calculated with the hypothesis contrast method with comparison of means for independent groups. In order to achieve an effect size with a confidence level that was set at 95% corresponding to an alpha value of 0.05 and a power of 80%, 6 patients per group are required and considering 20% losses, we will recruit 8 patients per group. group with a total of 24 patients.

Randomization: Study participants will be randomly assigned to one of the 3 exercise programs using a computer-generated hidden block randomization scheme (with Epidata software) with randomly varying blocks and stratification by sex (female or male), age (male or female). 18 to 44, 45 to 70 years), and AIS score (A, B, C or D). Participants will be assigned to their respective intervention according to the randomization schedule. Participants will be assigned a randomization number in the order they enroll.

Blinding: Those in charge of evaluating results and the person in charge of statistical analysis will be blinded and will not know the assignment of the intervention. The person in charge of carrying out the assigned exercise and the participant will know the assignment of the intervention.

Results analysis plan: For the analysis, a descriptive analysis is first proposed using measures of central tendency and dispersion for the quantitative variables and proportions for the qualitative variables. Analysis of variance will be performed to compare baseline characteristics between groups.

To know the distribution of the data, the Kolmogorov-Smirnov test will be carried out. Analysis of variance will be performed to compare the outcome measures at the end of training between the three groups.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of spinal cord injury with any American Spinal Injury Association Impairment Scale (AIS) classification
* Neurologic level below C8
* Time since injury greater than 6 months
* Any etiology
* Any type (complete and incomplete)
* Adequate trunk control (trunk control scale >13 points)

Exclusion Criteria:

* Another neurologic diagnosis
* Sense organ alteration
* Orthopedic problem that interferes with training
* Alteration in superior mental function
* Cardiovascular or metabolic disease that interferes with training

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 63 (Estimated)
Dates: Start 2023-01-25 (Actual); Primary Completion 2023-01-25 (Actual); Study Completion 2026-01-30 (Estimated)

PRIMARY OUTCOMES:
Measured metabolic equivalents | Before training and 8 weeks
  Metabolic unit of measurement that indicates the ml of oxygen consumed per kg/min
Oxygen consumption (VO2máx) | Before training and 8 weeks
  It is the largest amount of oxygen that the body can absorb, transport and consume in a given time.
Low-high frequency ratio (LF/HF) | Before training and 8 weeks
  Heart rate variability domain measurement

SECONDARY OUTCOMES:
Satisfaction with life | Before training and 8 weeks
  Life satisfaction questionnaire-9 is a validated questionnaire to assess life satisfaction in people with a spinal cord injury. It is composed of 9 questions that are rated by the patient between 1 (very dissatisfying) to 6 (very satisfying) and that explore perception in life as a hole, vocational, financial and leisure situations, contact with friends and acquaintances, sexual life and family life, partnership relation, physical and psychological health. Score ranges between 9 and 54. Higher values represent better results.
Spinal Cord Injury Independence Measure III | Before training and 8 weeks
  Validated specific independence measure for spinal cord injury. The main domains will be contemplated as secondary outcomes (Catz A, Spinal Cord 2007). Score ranges between 0 and 100. Higher values represent better results.
Plasma glucose concentration. | Before training and 8 weeks
  A blood glucose level less than 100 mg/dl was considered normal, values of 100-125 mg/dl were considered abnormal fasting blood glucose, and values greater than or equal to 126 mg/dl were considered diagnostic of diabetes mellitus.
Plasma triglyceride concentration | Before training and 8 weeks
  A concentration below 150 mg/dl was considered normal, higher concentrations were considered hypertriglyceridemia.
High-density lipoprotein cholesterol (HDL-C) | Before training and 8 weeks
  HDL cholesterol below a value of less than 40 mg/dl.
Low-density lipoprotein cholesterol | Before training and 8 weeks
  Elevated LDL cholesterol was defined as a value greater than or equal to 130 mg/dl.
Serum insulin | Before training and 8 weeks
  Serum insulin concentration in uU/ml determined by chemiluminescence
Ultrasensitive CRP | Before training and 8 weeks
  Serum CRP concentration mg/l
Appendicular lean mass to height ratio (ALM/Height2) | Before training and 8 weeks
  The amount of lean mass in the arms and legs relative to height.
Body mass index | Before training and 8 weeks
  Weight of a person in kilograms divided by the square of the height in meters in individuals
Trunk control Test | Before training and 8 weeks
  Score between 0-24, cut-off point 13. Higher values represent better results. The clinical trunk control test for individuals with spinal cord injury will be used

CONTACTS AND LOCATIONS:
Locations (1):
- Instituto Nacional de Rehabilitación "Luis Guillermo Ibarra Ibarra", Mexico City, Mexico City, Mexico

IPD SHARING:
Plan to Share IPD: Yes
Data base whithout identifications
Supporting Information: Study Protocol, SAP, ICF, Analytic Code
Time Frame: After January 2026 for 5 years
Access Criteria: Ask the authors directly by e-mail